CLINICAL TRIAL: NCT03571477
Title: Sleep Apnea : Diagnosis and Monitoring
Acronym: ApneaBand
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government); AIRFAN (Unknown); AGIR à Dom (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC18.010
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep apnea diagnosis; Sleep apnea monitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ApneaBand — Mesure of oxygen saturation (oximetry), pulse wave (photoplethysmography), electrodermal activity and movements (tri-axial accelerometer)

SUMMARY:
This prospective study aims to evaluate a new medical screening method to detect and discriminate sleep apnea-hypopnea events. A new device called ApneaBand will be tested to propose a new screening method facilitating the diagnosis and monitoring of the sleep apnea syndrom, still underdiagnosed. This device will be tested in comparison with polysomnography (PSG), the gold standard reference method of sleep apnea diagnosis.

DETAILED DESCRIPTION:
The objective of this study is to dertermine the performance of the ApneaBand, a new non-intrusive and portable device, in detecting sleep apnea, in comparison with PSG.

40 apneic and non apneic subjects will wear the ApneaBand recording the different sleep stages and the occurency of apnea-hypopnea sleep events through four sensors including oximetry (oxygen saturation), photoplethysmography (pulse wave), electrodermal activity and tri-axial accelerometer (movements).

Inclusion visit will be proceeded at the University Hospital Grenoble-Alpes ; polysomnography and mesures by the ApneaBand will be proceeded at the patient's home by IC@dom. Patients will be equiped with PSG + ApneaBand during the first night and with ApneaBand only the second night.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate or severe obstructive sleep apnea (OSA), diagnosed by polygraphy or PSG for less than 2 years, and not treated for that.
* Non apneic person (Berlin score = 0 or 1)
* Person be able to use the personal health monitoring device ApneaBand
* Be legally able to give consent
* Person affiliated to social security

Exclusion Criteria:

* Patient already treated for OSA
* Patient equipped with an electric medical device (non-exhaustive examples: cardiac pace maker, cochlear implant, neuro-stimulator)
* Being unable to understand and to follow recommendations for the study due to cognition or language problems
* Pregnant women, feeding and parturient
* Person under administrative or judicial control, or who is protected under the act
* Person in exclusion period for another study
* Person which would perceive more than 4500 euros of compensation because of its participation in other clinical studies in 12 months preceding this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with OSA and not treated for that
  * Non apneic subjects or unknown apneic subjects wishing to explore their sleep
  * Different skin tones from Fitzpatrick's phototypes I to VI.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Performance of the ApneaBand to detect sleep apnea | 3 days
  Performance of the ApneaBand device in detecting moderate to severe sleep apnea (defined by an Apnea-Hypopnea Index (AHI) ≥ 15 events/hour), in comparison with PSG

SECONDARY OUTCOMES:
Performance of the ApneaBand to mesure the apnea severity | 3 days
  Performance of the ApneaBand device in detecting sleep apnea according to its severity (2 pre-specified thresholds of AHI: > 5 and ≥ 30), in comparison with PSG
External reproductibility of AHI measurement by the ApneaBand | 3 days
  Reproducibility between AHI from polysomnography and ApneaBand
Internal reproductibility of AHI measurement by the ApneaBand | 3 days
  Reproducibility between different AHI mesures from ApneaBand
ApneaBand algorith validation for AHI measurement | 3 days
  External validation of the ApneaBand algorithm
Sleep stage detection by ApneaBand | 3 days
  To assess if electrodermal activity assessed by the ApneaBand during sleep is able to differerenciate the different sleep stages
Skin tone variability | 3 days
  To asses if oxygen saturation assessed by the ApneaBand could be performed in persons with dark skin tones

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Pr, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Chu Grenoble-Alpes, La Tronche, Isère, France